CLINICAL TRIAL: NCT01991704
Title: The Neural Mechanisms of the Incubation of Cue-induced Craving in Alcohol Dependence
Brief Title: Incubation of Alcohol Craving During Abstinence
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Dependence, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: nidd_peking
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Alcohol Dependence
Keywords: incubation; Craving; alcohol dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — The blood samples of all participants were collected at each point of withdrawal.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In order to determine whether the 'incubation of craving' phenomenon also occurred in alcoholics, investigators employed an experimental approach to investigate the time course of cue-induced craving in alcoholism. Eighty male participants were randomly divided into Four groups, and they were assessed at 7, 14, 30, and 60 days of abstinence for cue-induced alcohol craving . Another group including 19 patients was repeatedly tested for the cue-induced alcohol craving at the above abstinence days. Other psychological and physiological measures were administered at the four abstinence time points.

DETAILED DESCRIPTION:
All subjects provided written informed consent after a full explanation of the protocol design.

ELIGIBILITY:
Inclusion Criteria:

* met the criteria of DSM-IV for alcohol dependence
* aged 18-60 years,male

Exclusion Criteria:

* current or past history of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) axis I disorders
* with other serious physical diseases (respiratory disorders, cardiovascular disease and so on)
* other drug abuse except for nicotine

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: alcohol dependence
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
changes of alcohol craving measured with visual analogue scales | abstained from alcohol for 7 days, 14 days, 30 days and 60 days

SECONDARY OUTCOMES:
heart rate changes | 7, 14, 30 and 60 days after abstained
blood pressure changes in different abstinence days | 7, 14, 30 and 60 days after abstained
skin conductance changes in different abstinence days | 7, 14, 30 and 60 days after abstained
changes of Alcohol Urge Questionnaire | 7, 14, 30 and 60 days after abstained

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, Prof., Study Director — National Institute on Drug Dependence, China